CLINICAL TRIAL: NCT01122303
Title: Comparison of Corneal Epitheliotropic Factors in Autologous Serum Eye Drops Between Nonautoimmune Dry Eye and Stevens-Johnson Syndrome With Dry Eye
Brief Title: Corneal Epitheliotropic Factors in Autologous Serum Eye Drops in Nonautoimmune and Stevens-Johnson Syndrome With Dry Eye
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Pinnita Prabhasawat, Department of Ophthalmology, Faculty of Medicine Siriraj Hospital, Mahidol University
Other Study IDs: 520/2552(EC4)
Record Dates: First submitted 2010-05-01; First posted 2010-05-13 (Estimated); Last update posted 2010-05-13 (Estimated); Status verified 2010-05

CONDITIONS: Stevens-Johnson Syndrome
Keywords: Autologous serum eye drops; EGF; TGF-β1; TGF-β2; Fibronectin; Stevens-Johnson syndrome; Dry eye
MeSH Terms: conditions — Stevens-Johnson Syndrome; Dry Eye Syndromes

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SJS: Stevens-Johnson syndrome patients with dry eye
- Control: Non-autoimmune dry eye patients

SUMMARY:
Autologous serum eye drops (ASE) have been becoming popular in treatment of severe dry eye for the past decade. One of the most beneficial properties of the ASE over artificial eye drops is the epitheliotropic capacity owing to the presence of growth factors and other proteins. There have been reports on alteration of serum growth factors in autoimmune diseases such as rheumatoid arthritis. Alteration in serum growth factors may lead to different therapeutic effect of ASE. We therefore would like to know if there are any alteration growth factors, epidermal growth factor (EGF), transforming growth factor-beta1 (TGF-β1), transforming growth factor-beta2 (TGF-β2), and fibronectin, in ASE from Stevens-Johnson syndrome (SJS) patients with dry eye, which constitutes a major group of ASE usage in Siriraj Hospital, as compared with non-autoimmune dry eye. We also study stability of these factors following different storage conditions.

DETAILED DESCRIPTION:
Ten SJS patients with dry eye and 10 non-autoimmune dry eye patients are recruited in this study. Twenty to forty mL of peripheral venous blood is drawn and the serum is separated. The serum is diluted with Balanced Salt Solution (BSS) to provide 20% ASE. The levels of EFG, TGF-β1, TGF-β2, and fibronectin in 20% ASE are quantitated by enzyme-linked immunosorbent assay (ELISA) method and are compared between the two groups of samples. To study the stability of these serum factors under storage conditions used in clinical settings, 20% ASE are stored at different temperature and time i.e., at 4 ํC for 1 week and 1 month, and at -20 ํC for 1, 3 and 6 month. Their levels are then measured following each storage condition.

ELIGIBILITY:
Inclusion Criteria:

SJS group

* Patients diagnosed with SJS with dry eye syndrome
* Age more than 18 years old

Control group

* Patients diagnosed with dry eye syndrome
* Age more than 18 years old

Dry eye syndrome is defined as the having at least one symptom and one sign as the following:

Symptoms

1. Dryness sensation in the eye
2. Sandiness sensation in the eye
3. Burning sensation in the eye
4. Redness of the eye
5. Eye irritation
6. Eye stuck shut in the morning

Signs

1. Meibomian gland dysfunction
2. Tear film break-up time (TFBUT) < 10 sec
3. Fluorescein staining at cornea
4. Schirmer test without anesthesia score ≤ 5 mm / 5 min
5. Ocular surface problems

Exclusion Criteria:

* Taking immunosuppressive drugs
* Acquired immunodeficiency syndrome (AIDS) patients or other immunodeficiency conditions
* Having autoimmune disorders (except for SJS in case group)
* Having systemic underlying diseases such as uncontrolled diabetes mellitus (DM), chronic kidney disease, liver cirrhosis, or systemic infection
* Pregnant women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SJS patients with dry eye and non-autoimmune dry eye patients who are treated at Siriraj Hospital, Bangkok, Thailand
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-12; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Comparisons of the concentrations of EGF, TGF-β1, TGF-β2 and fibronectin in 20% ASE between SJS patients with dry eye and non-autoimmune dry eye patients | 1 year

SECONDARY OUTCOMES:
The concentrations EGF, TGF-β1, TGF-β2 and fibronectin in 20% ASE of SJS patients with dry eye syndrome and of non-autoimmune dry eye patients at different storage conditions i.e., at 4 °C for 1 week and 1 months, and at -20 °C for 1, 3 and 6 months | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pinnita Prabhasawat, MD, Principal Investigator — Department of Ophthalmology, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (1):
- Department of Ophthalmology, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand